CLINICAL TRIAL: NCT04755608
Title: The Effect OfF Low-Intensity Resistance Exercise Training Combined With Blood Flow Restruction On Triceps Brachii Muscle Volume And Performance
Brief Title: The Effect of Low-Intensity Resistance Exercise Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, Assist. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 46418926-19-138
Record Dates: First submitted 2021-01-30; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: muscle hypertrophy; triceps brachii; muscle strength

STUDY DESIGN:
Intervention Model Description: Self Controlled Randomised Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity Blood Flow Restriction Group (Experimental)
  Interventions: Other: Low Intensity Exercises with Blood Flow Restriction
- High Intensity Resistant Training Group (Active Comparator)
  Interventions: Other: High Intensity Resistant Exercise

INTERVENTIONS:
Other: Low Intensity Exercises with Blood Flow Restriction — In the exercise protocol, people exercised resistance between 20% and 30% of 1 MaxRepetition with free weight. In addition, blood flow was restricted in 70% of the arterial occlusion pressure of the individual with the help of a cuff during exercise.
  Arms: Low Intensity Blood Flow Restriction Group
Other: High Intensity Resistant Exercise — People included in the study did resistance exercise with free weight at 70-80% of 1 MT.
  Arms: High Intensity Resistant Training Group

SUMMARY:
It was to compare the effect of low-load resistance training with blood flow restriction (LL-BFR) and high-intensity resistance training (HI-RT) on muscle strength, endurance and volume, functional performance, and delayed onset muscle soreness (DOMS).

The study included 13 young women. It is a controlled study designed for individuals to perform two different exercise protocols unilaterally. The persons were randomly allocated into two groups as LI- BFR (Group I, n = 13) and HI-RT (Group II, n = 13). Both groups received training for 6 weeks and 3 days a week. Blood flow restriction was performed only in group I.

DETAILED DESCRIPTION:
Both sides triceps muscle thickness, triceps and biceps strength and endurance, functional performances (upper extremity Y balance test (UQYBT)), delayed-onset muscle soreness (DOMS) were evaluated before and after training.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-26,
* Do not have a chronic disease history and do not use medication,
* Female individuals were included.

Exclusion Criteria:

* People who made resisted exercise in the last 6 months,
* Smoker,
* BMI above 30 kg / m2,
* Individuals with hypertension were excluded.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Due to physiological differences between men and women, it was preferred to include only women.
Enrollment: 13 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
triceps muscle thickness | 6 weeks
  Triceps brachial (TB) long head thickness was measured using the Esaote mylab C series ultrasound device.
triceps and biceps strength | 6 weeks
  Triceps brachial muscle strength was evaluated with an isokinetic dynamometer (Cybex HUMAC / NORM, CSMI, 2004). Isometric muscle strength measurement was performed at the beginning and end of the study at angular velocities of 0-150 ° elbow range, 60 ° / s (strength measurement)
triceps and biceps endurance | 6 weeks
  Triceps brachial muscle strength was evaluated with an isokinetic dynamometer (Cybex HUMAC / NORM, CSMI, 2004). Isometric muscle strength measurement was performed at the beginning and end of the study at angular velocities of 0-150 ° elbow range, 180 ° / s (endurance measurement).
functional performances | 6 weeks
  Upper Extremity Y Balance Test
delayed-onset muscle soreness | 6 weeks
  Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Tütüneken, MSc, Principal Investigator — Istinye University
Locations (1):
- University and Health Sciences Physical Therapy and Rehabilitation, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No